CLINICAL TRIAL: NCT01167062
Title: Efficacy of Tamsulosin OCAS in the Conjunctive Medical Treatment of Distal Ureteral Stones.A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy of Tamsulosin Oral-controlled Absorption System (OCAS) in the Treatment of Distal Ureteral Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Bannakij Lojanapiwat M.D, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAM040-0109
Record Dates: First submitted 2010-07-16; First posted 2010-07-22 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-06

CONDITIONS: Ureteral Calculi
MeSH Terms: conditions — Ureteral Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Tamsulosin Hydrochloride OCAS 0.4 mg (Experimental)
  Interventions: Drug: Tamsulosin Hydrochloride OCAS 0.4 mg

INTERVENTIONS:
Drug: Tamsulosin Hydrochloride OCAS 0.4 mg — One tablet OD for a maximum of 28 days
  Arms: Tamsulosin Hydrochloride OCAS 0.4 mg
Other: Placebo — One tablet OD for a maximum of 28 days
  Arms: Placebo

SUMMARY:
This is a randomized double blind placebo-controlled study that will assess the efficacy of Tamsulosin oral-controlled absorption system (OCAS) 0.4 mg in the conjunctive medical treatment of distal ureteral stones with a size of 4-10 mm compared to placebo in control group.

DETAILED DESCRIPTION:
* patient will be randomized to receive placebo or Tamsulosin OCAS 0.4 mg 1 tablet OD for a maximum of 28 days or until the ureteral stone is passed and sodium diclofenac 50 mg twice a day, for 10 days.
* All patients will receive 75 mg sodium diclofenac via intramuscular on demand

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged => 18 years.
* Patients who have distal ureteral stones with a size of 4-10 mm
* Written informed consent has been obtained.

Exclusion Criteria:

* Patients with history of ureteral surgery
* Patients with urinary tract infection
* Patient with diabetes and peptic ulcer
* Patient with renal dysfunction (elevated of serum creatinine level)
* Patients with severe hydronephrosis
* Patients with history of passing stones
* Pregnancy
* Patients who desire to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Stone expulsion rate and time. | 28 days

SECONDARY OUTCOMES:
Number of diclofenac injection used | 28 days
Rate of occurrence of adverse events | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Maharat Nakhon Chiangmai Hospital, Muang, Chiangmai, Thailand